CLINICAL TRIAL: NCT05457569
Title: Acceptability and Feasibility of Implementing a Coordinated Hospital/Non-hospital Parenting Support and Prevention Program for Families of Infants at High Neurodevelopmental Risk After Neonatal Intensive Care Hospitalization
Acronym: PRéPaR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: JANDET ReSPIr 2021
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Neurodevelopmental Motor Disorders
MeSH Terms: interventions — Focus Groups; WP 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Parent Support Group - WP1: Group representatives (SOS Préma, The Neurogroup...)
  Interventions: Other: Focus group (FC) - WP1
- Parents of infants at a high risk of neurodevelopmental disorders - WP1: infants between 34 weeks' gestation and 4 months' corrected age at the time of the first focus group and with at least one risk factor for neurodevelopmental disorder
  Interventions: Other: Focus group (FC) - WP1
- Parents of children with developmental difficulties - WP1: children between 18 and 48 months corrected age at the time of the first focus group:
  * with at least one risk factor for neurodevelopmental disorder
  * presenting an abnormal, non-transient clinical state
  Interventions: Other: Focus group (FC) - WP1
- Health Professionals - WP1: Private physiotherapists, labor and delivery nurses of the Maternal and Child Protection, Centre d'action médico-sociale précoce (CAMSP) (psychomotricians, psychologists) and doctors involved in the care and follow up of children at risk of developmental disorders whose parents have agreed to participate in the study.
  Interventions: Other: Focus group (FC) - WP1
- Physiotherapist in a private practice - WP2: Physiotherapists working in a private practice
  Interventions: Other: Child Neurodevelopment Questionnaires - WP2; Other: Evaluation of compliance for the acquired skills in terms of development support - WP2; Other: Evaluation of physiotherapist satisfaction with the follow-up and the time spent at the consultation - WP2; Other: 4 Focus Group (FC) - WP2
- Parents - WP2: parents of hospitalized children between 34 weeks of gestation and 4 months of corrected age with at least one risk factor for neurodevelopmental disorder
  Interventions: Other: 4 Focus Group (FC) - WP2
- PMI-CAMPS - WP2: Labor and delivery nurses from the Protection Maternelle et Infantile, CAMPS (psychomotricians, psychologists) and doctors involved in the care of children at risk of developmental disorders who are in charge of the follow-up of children whose parents have agreed to participate in the study.
  Interventions: Other: 4 Focus Group (FC) - WP2

INTERVENTIONS:
Other: Focus group (FC) - WP1 — 3 group meetings for each group of parents:
  1. Parents only
  2. Parents and representatives of patient support groups
  3. Parents and health professionals specialized in the care of these children at risk
  Groups: Health Professionals - WP1; Parent Support Group - WP1; Parents of children with developmental difficulties - WP1; Parents of infants at a high risk of neurodevelopmental disorders - WP1
Other: Child Neurodevelopment Questionnaires - WP2 — during the 4th month of corrected infant age
  Groups: Physiotherapist in a private practice - WP2
Other: Evaluation of compliance for the acquired skills in terms of development support - WP2 — during the 4th month of corrected infant age
  Groups: Physiotherapist in a private practice - WP2
Other: Evaluation of physiotherapist satisfaction with the follow-up and the time spent at the consultation - WP2 — at the end of the study
  Groups: Physiotherapist in a private practice - WP2
Other: 4 Focus Group (FC) - WP2 — * Parents who accepted the follow-up
  * Parents who have partially completed the programme
  * Maternal and Child Protection & CAMSP professionals
  * Physiotherapists in a private practice
  Groups: PMI-CAMPS - WP2; Parents - WP2; Physiotherapist in a private practice - WP2

SUMMARY:
The PRéPaR project aims to construct, with the help of parents and early care providers, a support program for the families of infants at an increased risk for neurodevelopmental disorders, and to evaluate the acceptability and feasibility of such a program. This program aims to strengthen parenting skills, support infant development and improve the continuity of hospital/non-hospital care, including early identification of neurodevelopmental motor disorders and continuation of the support initiated during neonatal hospitalization.

ELIGIBILITY:
Inclusion Criteria:

WP1:

1. For the group of parents of children with documented neurodevelopmental difficulties, their child must meet the following three conditions:

   * Be between 18 months and 48 months corrected age at the time of the first focus group
   * Have at least one risk factor putting them at high neurodevelopmental risk at birth:

     * Preterm infant ≤ 31 WG + 6 days
     * Birth weight less than 1500g
     * Child who has had a stroke or stages 2 or 3 hypoxic-ischaemic encephalopathy of the newborn according to the Sarnat classification
     * Central neurological lesion, diagnosed on brain imaging.
   * Present an abnormal, non-transient clinical state: diagnosis of cerebral palsy made or in progress (GMFCS 1 to 5), central neurological syndrome, diagnosed neurodevelopmental disorder.

   The parents must be able to participate in the 3 interviews (T1, T2 and T3).
2. For the group of infants at high neurodevelopmental risk at hospital discharge, their child must meet the following two conditions:

   * Be between 34 weeks of amenorrhea (i.e., 1.5 months premature) and 12 months of corrected age at the time of the first focus group,
   * Have at least one risk factor putting them at high neurodevelopmental risk at birth:

     * Preterm infant ≤ 31 WG + 6 days
     * Birth weight less than 1500g
     * Child who has had a stroke or stages 2 or 3 hypoxic-ischaemic encephalopathy of the newborn according to the Sarnat classification
     * Central neurological lesion, diagnosed on brain imaging.

   The parents must be able to participate in the 3 interviews (T1, T2 and T3).
3. Professionals and parent support groups:

Physiotherapists in private practice, labor and delivery nurses of the Maternal and Child Protection, CAMSP (psychomotricians, psychologists) and doctors involved in the care of children at developmental risk in charge of the follow-up of children for whom the parents have agreed to participate in the study. These professionals must in turn have agreed to participate in the study. User representatives (SOS Préma, Le Neurogroup...) who have agreed to participate in the study.

WP2:

1. Parents of children hospitalized in the neonatal services of the CHU Dijon who meet at least one of the following criteria:

   * Be between 34 weeks of amenorrhea (1.5 months premature) and 3 months of corrected age (3 months post-term)
   * Have at least one risk factor putting them at high neurodevelopmental risk at birth:

     * Child who has had a stroke or stages 2 or 3 hypoxic-ischaemic encephalopathy of the newborn according to the Sarnat classification
     * Central neurological lesion, diagnosed on brain imaging.
2. Professionals:

Physiotherapists in private practice, labor and delievery nurses of the Maternal and Child Protection, CAMSP (psychomotricians, psychologists) and physicians involved in the care of children at developmental risk in charge of the follow-up of the children whose parents agreed to participate in the study. These professionals must in turn have agreed to participate in the study.

Exclusion Criteria:

* Parents who are physically or cognitively unable to participate in a group interview or who do not have a sufficient command of French.
* Parents who are minors
* Parents under legal protection
* Parents of children with major orthopedic or traumatic disorders unrelated to the high risk of cerebral palsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of infants at high risk of neurodevelopmental disorders Parents of children with developmental disorders
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Typology, categorization and operationalization of parental needs and expectations | Through WP1 completion an average of 18 months
  These will be used to develop of the early education program
Typology of perceived subjective representations and description of barriers and levers to use with parents and professionals | through WP2 completion an average of 16 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France